CLINICAL TRIAL: NCT07313319
Title: Trial of Underwater Birth: A Randomized Control Trial
Brief Title: Trial of Underwater Birth
Acronym: TUB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-454; Lacks Grant (Other: University of New Mexico)
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Birth
Keywords: waterbirth; landbirth; epidural use; birth outcomes
MeSH Terms: interventions — Natural Childbirth

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Land Birth (No Intervention): Study subjects enrolled in the land birth cohort of this study will receive care as usual on labor and delivery. There will be no changes to their intrapartum care including their ability to use water as a form of pain relief during labor (Stage 1 water immersion) if deemed appropriate by their care team. Land birth participants who use water for pain relief will be assisted out of the water prior to second stage (pushing) as is currently routine on UNMH Labor and Delivery.
- Waterbirth (Experimental): Subjects enrolled in the waterbirth cohort will be assessed for continued eligibility at time of admission to labor and delivery and continuously during labor. Those who remain eligible will have an inflatable birthing tub set up in their room and available for them to use as desired. Waterbirth will be performed in adherence to the following protocol endorsed by the American College of Nurse Midwives.
  Interventions: Procedure: Waterbirth

INTERVENTIONS:
Procedure: Waterbirth — Those who remain eligible will have an inflatable birthing tub set up in their room and available for them to use as desired. Waterbirth will be performed in adherence to the following protocol endorsed by the American College of Nurse Midwives.
  Arms: Waterbirth

SUMMARY:
Evaluate maternal perinatal outcomes in adult low-risk laboring people randomized to waterbirth compared to those randomized to birth on land.

DETAILED DESCRIPTION:
The proposed randomized control trial will be approached as a pilot study to explore or test (if sample size permits) our hypotheses.

Primary outcome: Use of epidural anesthesia during labor and vaginal birth.

Secondary outcomes: Use of IV narcotics in labor, duration of active labor, mode of delivery, composite maternal adverse outcomes (see below), use of intermittent auscultation (IA), composite neonatal adverse outcomes (see below), United States Birth Satisfaction Scale-Revised (US-BSS-R), use of epidural analgesia during labor (full intention-to-treat analysis).

ELIGIBILITY:
Inclusion Criteria: Inclusion criteria based on A model practice template for hydrotherapy in labor and birth (2016):

Prenatal inclusion criteria (to be assessed at the time of enrollment):

* ≥18 years of age
* Able to speak and understand English or Spanish
* Singleton gestation
* Vertex presentation
* Able to ambulate with no mobility restrictions (i.e., no difficulty getting from seated to standing)
* Less than class III obesity (BMI <40 kg/m2) at initiation of prenatal care

Labor inclusion criteria (to be assessed at time of admission):

* Greater than 37 weeks 0 days through and less than 412 completed weeks 6 days gestation with fetus in vertex presentation
* Normal blood pressure and normal temperature (obstetric criteria for exclusion: two blood pressures 140/90 four hours apart; two fevers of over 100.4 one hour apart)

Exclusion Criteria: based on A model practice template for hydrotherapy in labor and birth (2016):

Prenatal exclusion criteria (to be assessed at the time of enrollment):

* Active infections such as HIV, Hepatitis B, Hepatitis C, HSV outbreak (on prophylaxis acceptable) (GBS positive is acceptable)
* Pre-existing medical conditions including heart disease, uncontrolled asthma, preexisting diabetes, chronic hypertension, or activity restrictions
* High-risk pregnancy conditions including preeclampsia, gestational hypertension, preterm gestation, multiple gestation, gestational diabetes type A2, estimated fetal weight of 5000g for non-diabetics or >4500 for GDM-A1, unstable substance use disorder (i.e. not in remission), placental abruption or other unexplained vaginal bleeding, previous cesarean section, fetal growth restriction (<10th percentile), fetal anomaly, or other neonatal condition that may complicate neonatal transition to extrauterine life.
* Existing contraindication to vaginal birth

Labor exclusion criteria (to be assessed at the time of admission):

* Meconium-stained amniotic fluid
* Preterm rupture of membranes (PROM) greater than 24 hours without the start of any labor contractions (those whose have PROM greater than 24 hours but are in labor can continue to be included in the study)
* Immediate need for operative delivery at time of admission

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Epidural Anesthesia | Labor and delivery
  Evaluate the epidural anesthesia rate in adult low-risk laboring people randomized to have the option of waterbirth compared to those randomized to birth on land.

SECONDARY OUTCOMES:
IV Narcotic Use | Labor and delivery
  Use of IV narcotics in labor
Active Labor Duration | Labor and delivery
  duration of active labor
Delivery Mode | Labor and delivery
  Mode of delivery
Maternal Adverse Outcomes | Up to 2 weeks postpartum
  Composite maternal adverse outcomes
Intermittent Auscultation (IA) | Labor and delivery
  Use of intermittent auscultation (IA)
Neonatal Adverse Outcomes | Up to 2 weeks postpartum
  Composite neonatal adverse outcomes
United States Birth Satisfaction Scale-Revised (US-BSS-R) | 3 days to 2 weeks postpartum
  Satisfaction with birth experience

CONTACTS AND LOCATIONS:
Overall Officials: Katrina Nardini, Principal Investigator — University of New Mexico